CLINICAL TRIAL: NCT05637359
Title: Tracked Ultrasound for Patient Registration in Surgical Navigation During Abdominal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRBd20-141
Record Dates: First submitted 2022-09-08; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Abdominal Cancer
Keywords: Surgical Navigation; Ultrasound; Registration; Electromagnetic Tracking; Pelvic Malignancies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients scheduled for navigated abdominal cancer surgery: Patients are 18 years old or older. Patients are scheduled for tumor surgery in the abdominal/pelvic area and navigation surgery with a scheduled Cone Beam CT-scan in the operating room. Patients provide written 'informed consent'. The to be administered intervention is a percutaneous tracked ultrasound measurement of the patient's pelvic bone on the operating room after anesthesia.
  Interventions: Device: Tracked ultrasound measurement

INTERVENTIONS:
Device: Tracked ultrasound measurement — Participation in the study will not involve additional visits to the hospital or additional CT scans for the included patients. For this experiment, 2D ultrasound images are obtained using an ultrasound transducer linked to the electromagnetic navigation system, which is already in place for the navigation at the operating room. After anesthesia and in parallel to the final preparations of the patient, two percutaneous ultrasound measurements of the pelvic bone are performed and recorded. The first measurements are performed in Trendelenburg patient position and the second measurements in supine patient position. When preparations are finished, normal workflow is continued, including the standard Cone Beam CT acquisition required for the navigation and sterile draping of the patient.
  The acquired ultrasound scans will be analyzed post-operatively and offline. This measurement has no impact on the (navigated) surgical procedure itself.

SUMMARY:
The goal of this observational pilot study is to evaluate the feasibility and accuracy of tracked ultrasound registration on patients undergoing abdominal cancer navigation surgery. The main research question is: Could tracked ultrasound be applied as an alternative to standard CBCT scanning in surgical navigation? Participants will undergo tracked ultrasound measurements of the pelvic bone on the operating room after patient anesthesia and before surgical incision.

DETAILED DESCRIPTION:
Image-guided navigation surgery allows for full utilization of pre-operative imaging during surgery and has the potential of reducing both irradical resections and morbidity. Currently, registration is done by Cone-Beam CT (CBCT) scanning on the operating room (OR) prior to navigation surgery. However, standard CBCT scanning has several limitations, mainly limited availability on the hybrid OR and radiation exposure. Furthermore, standard CBCT scanning can only be performed in horizontal patient position, while the patient position mostly differs during surgery, such as the Trendelenburg position. The use of tracked ultrasound instead of standard CBCT could overcome these limitations, which might lead to an increased navigation accuracy and improved surgical outcomes. Therefore, the goal of this research is to evaluate the feasibility and accuracy of tracked ultrasound registration on patients undergoing abdominal cancer navigation surgery. The main research question is: Could tracked ultrasound be applied as an alternative to standard CBCT scanning in surgical navigation?

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients scheduled for tumor surgery in the abdominal/pelvic area and navigation surgery with a scheduled CBCT-scan in the OR
* Patients provide written 'informed consent'

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cancer in the pelvic-abdominal area, who are scheduled for surgical resection of the malignant tissue in combination with the surgical navigation technique.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Accuracy of tracked ultrasound registration. | One day
  To evaluate the accuracy of tracked ultrasound registration on patients undergoing abdominal cancer navigation surgery. This will be assessed using the target registration error in mm, where a lower error means a better outcome.

SECONDARY OUTCOMES:
Influence of patient position alteration on registration accuracy. | One day
  What is the influence of patient position alteration on the surgical navigation accuracy for standard Cone Beam CT and tracked ultrasound registration methods? This will be assessed using the target registration discrepancy in mm.
Measurement time of tracked ultrasound registration. | One day
  The time duration of ultrasound measurements will be recorded and compared with the conventional Cone Beam CT method. A faster ultrasound measurement time means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Theo Ruers, prof. dr., Principal Investigator — NKI
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hiep MAJ, Heerink WJ, Groen HC, Ruers TJM. Feasibility of tracked ultrasound registration for pelvic-abdominal tumor navigation: a patient study. Int J Comput Assist Radiol Surg. 2023 Sep;18(9):1725-1734. doi: 10.1007/s11548-023-02937-8. Epub 2023 May 25. PMID 37227572